CLINICAL TRIAL: NCT04918199
Title: Computer Based, vs Human Based Assessment of Kidney Allograft Failure Prediction and Stratification
Brief Title: Human Versus Computer-based Predictions of Long Allograft Survival
Acronym: iBox vs Human
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: iBoxvsHuman
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplant Failure
Keywords: iBox; individual risk prediction; kidney transplantation; long-term allograft outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paris Transplant Group cohort: 400 (10%) of the patients were randomly selected from 4,000 consecutive patients over 18 years of age prospectively enrolled at the time of kidney transplantation from a living or deceased donor at Necker Hospital, Saint-Louis Hospital, Foch Hospital, and Toulouse Hospital between January 1, 2005, and January 1, 2014, in France.
  Interventions: Device: Computer based assessment (iBox); Other: Physician assessement

INTERVENTIONS:
Device: Computer based assessment (iBox) — Individual allograft survival probabilities of death censored allograft survival seven years after the time of risk evaluation, computed using the iBox (NCT03474003), a qualified prognostication system designed to predict long term allograft survival up to seven years after evaluation.
Other: Physician assessement — Based on anonymized electronic health records, physicians have to determine a percentage of death censored allograft survival seven years after the time of risk evaluation,

SUMMARY:
The clinical decision-making after kidney transplantation is mainly driven by patient individual assessment. However, this task remains difficult and uncertain due to the integration of complex and numerous parameters. We aim to evaluate and compare the ability of transplant physicians to predict long term allograft survival compared with a computer-based survival prediction algorithm (iBox system).

DETAILED DESCRIPTION:
400 kidney transplant recipients among the cohort of 4,000 patients from the Paris Transplant Group prospective kidney transplant cohort (NCT03474003) were randomly selected. We generated an anonymized electronic health record for each included patient including a total of 60 classical kidney transplant prognostic parameters comprising baseline transplant and recipient characteristics, together with post-transplant parameters including allograft function, proteinuria, histology, diagnoses, and immunological profile collected during the first-year post-transplant. The time of risk evaluation for the human and the iBox system were at 1-year post transplant and the death censored allograft survival predictions made at 7 years after risk assessment. We enrolled transplant physicians at various stages of their careers (residents, fellows and seniors) to assign death censored graft survival probabilities at 7 years post risk assessment. The physicians were blinded to the actual patient outcome (allograft failure) and the iBox predictions. The physicians-based predictions will then be compared with the iBox system, a validated computer-based kidney survival prediction system.

ELIGIBILITY:
Inclusion Criteria:

* transplant evaluation available at one year post-transplant

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 (10%) of the patients were randomly selected with an evaluation available at one-year post-transplant from the Paris Transplant Group cohort, which gathers 4,000 consecutive patients over 18 years of age prospectively enrolled at the time of kidney transplantation from a living or deceased donor at Necker Hospital, Saint-Louis Hospital, Foch Hospital, and Toulouse Hospital between January 1, 2005, and January 1, 2014, in France.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Death censored allograft failure seven years after risk assessment | 7 years
  Predictions performances to predict allograft failure defined as a patient's definitive return to dialysis or preemptive kidney retransplantation after risk assessment.

SECONDARY OUTCOMES:
Evaluation of the parameters' importance in the prediction for physicians | 7 years
  Mean decrease in accuracy from a random survival forest from each physician will be used to determine the relative importance of the first ten parameters that led to their predictions.
Inter-rater agreement | 7 years
  Fleiss kappa will be used to measure inter-rater agreement between each physician's ranking

CONTACTS AND LOCATIONS:
Locations (1):
- Paris Translational Centre for Organ Transplantation, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loupy A, Aubert O, Orandi BJ, Naesens M, Bouatou Y, Raynaud M, Divard G, Jackson AM, Viglietti D, Giral M, Kamar N, Thaunat O, Morelon E, Delahousse M, Kuypers D, Hertig A, Rondeau E, Bailly E, Eskandary F, Bohmig G, Gupta G, Glotz D, Legendre C, Montgomery RA, Stegall MD, Empana JP, Jouven X, Segev DL, Lefaucheur C. Prediction system for risk of allograft loss in patients receiving kidney transplants: international derivation and validation study. BMJ. 2019 Sep 17;366:l4923. doi: 10.1136/bmj.l4923. PMID 31530561